CLINICAL TRIAL: NCT06757855
Title: A Multicenter, Single-arm I/II Clinical Study of Olverembatinib Combined With Venetoclax and Azacitidine in in Blast Phase Ph Chromosome- Chronic Myeloid Leukemia
Brief Title: Olverembatinib Combined With Venetoclax and Azacitidine in Blast Phase Ph Chromosome-positive CML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024090
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-12

CONDITIONS: CML,Blast Phase
MeSH Terms: interventions — olverembatinib; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olverembatinib Combined With Venetoclax and Azacitidine (Other)
  Interventions: Drug: Olverembatinib; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Olverembatinib — induction therapy：40mg,QOD；
  consolidation maintenance therapy: If patients with CMR are reduced to 30mg.
Drug: Venetoclax — induction therapy：leverl 0: 100mg d-2; 200mg d-1; 400mg d1-14
  leverl -1: 100mg d-2; 200mg d-1; 400mg d1-7
  leverl 1: 100mg d-2; 200mg d-1; 400mg d1-21
  consolidation maintenance therapy: 400mg d1-7
Drug: Azacitidine — induction therapy：75mg/m2/d, d1-7
  consolidation maintenance therapy: 75mg/m2/d, d1-7

SUMMARY:
Even in the TKI era, the outcoms of patients with blast phase is still poor.The response rate to conventional intensive chemotherapy is only 12.5% and the 5-year survival rate is 0 for patients with myeloid blast crsis. The response rate of TKI monotherapy is about 50% and the response rate is further improved when combined TKI and chemotherapy for patients with lymphoid blast crsis. The induction remission rate of chemotherapy alone for patients with Ph-positive acute lymphoblastic leukemia is 50-60%, and the remission rate increases to more than 95% when combined with TKI. Therefore, the application of TKI for patients in the blast crisis phase is of great significance. Olverembatinib is the only third-generation TKI drug approved in the Chinese mainland at present. Preclinical research data show that olverembatinib has a significant inhibitory effect on wild-type and mutant ABL resistant to the first and second-generation TKIs, as well as some complex mutations resistant to ponatinib. Phase I and II clinical studies have shown that for CML patients in the chronic and accelerated phases with resistance or intolerance to various TKIs, with or without T315I mutations, there are significant hematological and molecular responses and survival benefits. Olverembatinib can also inhibit many other kinases related to tumors. In vitro studies have shown that olverembatinib downregulates MCL-1 expression and acts synergistically with BCL-2 inhibitors to induce apoptosis of AML cells.

Preclinical studies have shown that venetoclax has a synergistic effect with TKIs. It upregulates apoptosis-inducing proteins, downregulates anti-apoptotic protein MCL1, inhibits the anti-apoptotic activity of BCL-XL, induces apoptosis of Ph+ cells, overcomes TKI resistance, and eliminates CML leukemia stem cells.

A large amount of evidence indicates that DNA hypermethylation plays an important role in the progression of CML, and abnormal DNA methylation is associated with progression to the accelerated and blast crisis phases and resistance to TKIs.Domestic scholars have reported successful cases of combined treatment with TKI, venetoclax, and demethylating agent azacitidine for CML patients with lymphoid blast crisis.

Therefore, we designed this study to explore the efficacy and safety of olverembatinib, venetoclax, and azacitidine in the treatment of CML patients in the blast crisis phase.

DETAILED DESCRIPTION:
In patients with chronic myeloid leukemia (CML) in the blase crsis phase who are aged≥15 years, olverembatinib combined with venetoclax and azacitidine was applied for induction and consolidation therapy. After remission, allogeneic stem cell transplantation was performed or olverembatinib combined with venetoclax and azacitidine was continued for consolidation and maintenance therapy. The maximum tolerated dose of the combined chemotherapy of olverembatinib, venetoclax and azacitidine was determined, and the efficacy and safety of the combined chemotherapy were evaluated.

Primary Endpoints Phase I: Determine the maximum tolerated dose of the combined chemotherapy of olverembatinib, venetoclax and azacitidine.

Phase II: Determine the complete hematological response rate (CHR) after 2 courses of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with t(9;22)(q34;q11)/BCR::ABL1 positive blast-phase CML who are aged 15 years or older, whether initially in the blast phase or progressing from the chronic phase, with no gender restriction.

   Blast phase criteria: Conforming to the 2022 WHO criteria for CML Blast phase: bone marrow or peripheral blood blast cells ≥ 20%; for diagnosis of acute lymphoblastic transformation, if the immature lymphoblasts (determined by immunophenotype) ≥ 5% according to the ICC 2022 criteria; blast cell aggregation in bone marrow or extramedullary tissues.
2. ECOG performance status score ≤ 2.
3. Major organ function assessment criteria: Total bilirubin < 1.5×upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN; serum creatinine < 2×ULN; myocardial enzymes < 2×ULN; serum amylase ≤ 1.5×ULN; left ventricular ejection fraction (LEF) within the normal range on echocardiography.
4. Men and women of reproductive potential agree and adopt effective contraceptive measures.
5. The informed consent form is signed by the patient himself/herself or an immediate family member. Considering the patient's condition, if the patient's signature is not conducive to the control of the disease, the legal guardian or an immediate family member of the patient signs the informed consent form.

Exclusion Criteria:

1. Before group entry, other systemic anti-cancer treatments for acute transformation were received (excluding single-agent TKI, hormone, or hydroxyurea for reducing tumor burden before group entry, and single-agent olverembatinib ≤ 14 days)
2. Myocardial infarction occurred within 12 months before enrollment in this study; other clinically significant cardiac diseases (such as unstable angina, congestive heart failure, uncontrollable hypertension, uncontrollable arrhythmia, etc.)
3. Uncontrolled active severe infection
4. Known positive serum HIV
5. Acute pancreatitis occurred within 1 year before study screening, or a history of chronic pancreatitis
6. Uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL, i.e., 5.1 mmol/L) or hypercholesterolemia (total cholesterol (TC) ≥ 6.2 mmol/L)
7. Another malignancy diagnosed and treated within 5 years before diagnosis, or previously diagnosed with another malignancy with evidence of residual disease. Patients with non-melanoma skin cancer or any type of carcinoma in situ, if completely resected, should not be excluded
8. Pregnant or lactating women
9. Clinical manifestations of CNS leukemia or extramedullary infiltration
10. Uncontrolled diabetes, defined as glycated hemoglobin value > 7.5%. Patients with previously existing but well-controlled diabetes need not be excluded
11. Mental illness that may prevent the subject from completing treatment or providing informed consent
12. Other conditions considered unsuitable for this study by the investigator

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-01-26 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of combination with olverembatinib, venetoclax and azacitidine | six weeks from day 1 of each course
  The standard "3+3" method is used to determine the maximum tolerated dose. There are 3 dose groups.
Determine complete hematological response rate (CHR) after 2 courses | six weeks after day 1 of 2nd courses of the treatment
  CHR is one of the evaluation criteria of treatment.

SECONDARY OUTCOMES:
Partial Cytogenetic Response（PCyR） | up to 2 years
  PCyR is an important clinical indicator for determining whether patients with CML are responding well to the treatment they are receiving.
Complete Cytogenetic Response（CCyR） | up to 2 years
  It is another important indicator used to assess the response to treatment in patients with chronic myeloid leukemia (CML). In the CCyR state, the patient's bone marrow cells no longer detect any abnormal cells carrying the Philadelphia chromosome.
Major Molecular Response（MMR） | up to 2 years
  When the test results show that the expression level of the BCR-ABL gene is reduced below a specific threshold, the patient is considered to have achieved MMR.
Deep Molecular Response（DMR） | up to 2 years
  It is an advanced indicator to assess the response of patients with chronic myeloid leukemia (CML) to treatment. DMR indicates that the expression level of the BCR-ABL fusion gene has been reduced to a very low level, which usually indicates that the patient's disease is in a very stable controlled state with a low risk of recurrence.
overall survival (OS) | up to 2 years after the date of the last enrolled participants
  Used to evaluate all patients who enter clinical trials. From the date of entry into the trial until the date of patient death (including any cause) or last survival follow-up.
Relapse-free survival (RFS) | up to 2 years after the date of the last enrolled participants
  Defined only for patients achieving CRc; measured from the date of achievement of remission until the date of hematologic relapse or death from any cause; patients not known to have relapsed or died at last follow-up are censored on the date they were last known to be alive
Therapeutic toxicity | up to 2 years after the date of the last enrolled participants
  This is a safety indicator and focuses on treatment-related toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No